CLINICAL TRIAL: NCT01647542
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, 24-week Study to Evaluate the Efficacy and Safety of Daily Oral TAK-875 25 and 50mg Compared With Placebo in Asia Pacific Subjects With Type 2 Diabetes
Brief Title: Study to Evaluate the Efficacy and Safety of Daily Oral TAK-875 25 and 50mg in Asia Pacific Adults With Type 2 Diabetes
Acronym: GRAND-307
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to potential concerns about liver safety (See Detailed Description)
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-875_307; U1111-1129-7865 (Registry Identifier: WHO); 1015011378 (Registry Identifier: TCTIN (Taiwan))
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Results first posted 2015-08-19 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Drug therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — TAK-875

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TAK-875 25 mg (Experimental): TAK-875 25 mg tablets, orally, once daily for up to 24 weeks.
  Interventions: Drug: TAK-875
- TAK-875 50 mg (Experimental): TAK-875 50 mg tablets, orally, once daily for up to 24 weeks.
  Interventions: Drug: TAK-875
- Placebo (Placebo Comparator): TAK-875 placebo-matching tablets, orally, once daily for up to 24 weeks.
  Interventions: Drug: TAK-875 Placebo

INTERVENTIONS:
Drug: TAK-875 — TAK-875 tablets
  Arms: TAK-875 25 mg; TAK-875 50 mg
Drug: TAK-875 Placebo — TAK-875 placebo-matching tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of TAK-875 in Asia Pacific adults with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-875. TAK-875 is being tested to treat people who have diabetes.

The study will enroll approximately 750 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* TAK-875 25 mg once daily
* TAK-875 50 mg once daily
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient

All participants will be asked to take one tablet at the same time each day throughout the study. All participants will be asked to record any time they have low blood sugar symptoms in a diary.

This multi-centre trial will be conducted the Asia Pacific region. The overall time to participate in this study is 30 weeks. Participants will make 13 visits to the clinic.

Due to potential concerns about liver safety, on balance, the benefits of treating patients with fasiglifam (TAK-875) do not outweigh the potential risks.

For this reason, Takeda has decided voluntarily to terminate the development activities for fasiglifam.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the patient is capable of understanding and complying with protocol requirements.
2. The patient or, when applicable, the patient's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Male or female, aged at least 18 years or over the legal age of consent in countries where that is greater than 18 years, with a historical diagnosis of T2DM.
4. Has an HbA1c of 7.0% to 10.0%, inclusive at screening, and has been treated with diet and exercise for at least 3 months.
5. Has a body mass index (BMI) of ≤45 kg/m^2 at screening.
6. Patients regularly using, non-excluded medications, must be on a stable dose for at least 4 weeks prior to Screening. However, PRN (as needed) use of prescription or over-the-counter medication is allowed at the discretion of the investigator.
7. A female of childbearing potential who is sexually active with a nonsterilized male partner agrees to routinely use adequate contraception from signing of the informed consent throughout the duration of the study and for 30 days after the last dose of study drug.
8. Is able and willing to monitor glucose with a home glucose monitor and consistently record his or her own blood glucose concentrations and complete subject diaries.

Exclusion Criteria:

1. Is unable to understand the official language (verbal or written) of the country for which a certified translation of the approved informed consent is available.
2. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, or sibling; biological or legally adopted) or may consent under duress.
3. Has hemoglobin a level ≤12 g/dL (≤120 g/L) (males) and ≤10 g/dL (≤100 g/L) (females) at the Screening Visit.
4. Has a history of any hemoglobinopathy that may affect determination of HbA1c.
5. Donated or received any blood products within 12 weeks prior to Screening or is planning to donate blood during the study.
6. Has systolic blood pressure ≥160 mm Hg or diastolic pressure ≥95 mm Hg at Screening or Baseline (If the patient meets this exclusion criterion, the assessment may be repeated once at least 30 minutes after initial measurement and decision will be made based on the second measurement).
7. Had coronary angioplasty, coronary stent placement, coronary bypass surgery, myocardial infarction, unstable angina pectoris, clinically significant abnormal electrocardiogram, cerebrovascular accident or transient ischemic attack within 3 months prior or at Screening.
8. Has a serum creatinine level of ≥1.5 mg/dL (males) and ≥1.4 mg/dL (females) and/or estimated glomerular filtration rate (GFR) <60 mL/min/1.73m^2 at Screening.
9. Has uncontrolled thyroid disease.
10. Has a history of laser treatment for proliferative diabetic retinopathy within 6 months prior to Screening.
11. Has a history or treatment for diabetic gastric paresis, gastric banding, or gastric bypass surgery.
12. Has alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) levels >2.0x the upper limit of normal range (ULN) at Screening.
13. Has a total bilirubin level greater than the ULN at Screening. Exception: if a patient has documented Gilbert's Syndrome, they will be allowed with an elevated bilirubin level per the investigator's discretion.
14. Has a known history of infection with human immunodeficiency virus (HIV), Hepatitis B virus (HBV), or Hepatitis C virus (HCV).
15. If a patient has no known history of HBV infection, then a HBV Screening test panel should be done. If the test is positive and there is clinical manifestation of active infection per Investigator's diagnosis, then the patient should be excluded. In addition, if the patient is considered to need antiviral treatment, the patient should be excluded. (If the test results indicate only an hepatitis B surface antigen (HBsAg) carrier without any clinical manifestation of active infection, and no antiviral treatment is needed, then the patient could be enrolled provided all other criteria are met.)
16. Has a history of cancer that has been in remission for <5 years prior to Screening. A history of basal cell carcinoma or stage 1 squamous cell carcinoma of the skin is allowed.
17. Has received any investigational compound within 30 days prior to Screening or has received >7 days of any antidiabetic agent within 3 months prior to Screening.
18. Has received TAK-875 in a previous clinical study.
19. Has a history of hypersensitivity, allergies or has had an anaphylactic reaction(s) to any component of TAK-875.
20. Has a history of drug abuse (defined as illicit drug use) or a history of alcohol abuse (defined as regular or daily consumption of more than 4 alcoholic drinks per day) within 2 years prior to Screening.
21. Received excluded medications prior to Screening or is expected to receive excluded medications.
22. If female, is pregnant (confirmed by laboratory testing, ie, serum/urine human chorionic gonadotropin (hCG), in females of childbearing potential) or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
23. If male, intends to donate sperm during the course of this study or for 30 days after final study medication dose.
24. Has any other physical or psychiatric disease or condition that in the judgment of the investigator may affect life expectancy or may make it difficult to successfully manage and follow the subject according to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2012-10; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (51):
- Australia (5):
  - Brookvale, New South Wales
  - Maroubra, New South Wales
  - Mosman, New South Wales
  - Woy Woy, New South Wales
  - Elizabeth Vale, South Australia
- China (30):
  - Hefei, Anhui
  - Beijing, Beijing Municipality
  - Beijing,P.R., Beijing Municipality
  - Chongqing, Chongqing Municipality
  - Fuzhou, Fujian
  - Xiamen, Fujian
  - Guangzhou, Guangdong
  - Guiyang, Guizhou
  - Shijiazhuang, Hebei
  - Harbin, Heilongjiang
  - Wuhan, Hubei
  - Changsha, Hunan
  - Chenzhou, Hunan
  - Nanjing, Jiangsu
  - Suzhou, Jiangsu
  - Changchun, Jilin
  - Changchun City, Jilin Province, Jilin
  - Xi'an, Shaanxi
  - Shanghai, Shanghai Municipality
  - Xi’an, Shanxi
  - Chengdu, Sichuan
  - Tianjin, Tianjin Municipality
  - Beijing
  - Chongqing
  - Guangzhou
  - Guiyang
  - Heilongjiang
  - Nanjing
  - Shanghai
  - Tianjin
- New Zealand (5):
  - Auckland
  - Hamilton
  - Rotorua
  - Tauranga
  - Wellington
- South Korea (6):
  - Goyang-si, Gyeonggi-do
  - Seongnam-si, Gyeonggi-do
  - Suwon, Gyeonggi-do
  - Gyeonggi-do
  - Incheon
  - Seoul
- Taiwan (5):
  - Kaohsiung City
  - New Taipei City
  - Taichung
  - Tainan
  - Taipei

REFERENCES:
- [Derived] Shavadia JS, Sharma A, Gu X, Neaton J, DeLeve L, Holmes D, Home P, Eckel RH, Watkins PB, Granger CB. Determination of fasiglifam-induced liver toxicity: Insights from the data monitoring committee of the fasiglifam clinical trials program. Clin Trials. 2019 Jun;16(3):253-262. doi: 10.1177/1740774519836766. Epub 2019 Mar 18. PMID 30880443

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 59 investigative sites in Australia, China, the Republic of Korea, New Zealand and Taiwan from 30 July 2012 to 18 March 2014.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus (T2DM) who were inadequately controlled when treated with only diet, exercise and any antidiabetic agent for less than or equal to (<=) 7 days within 12 weeks prior to Screening, were enrolled in 1 of 3 treatment groups: placebo; fasiglifam 25 milligram (mg); fasiglifam 50 mg.
Groups:
- Placebo: Fasiglifam placebo-matching tablets, orally, once daily, for up to 24 weeks.
- Fasiglifam 25 mg: Fasiglifam 25 mg, tablets, orally, once daily, for up to 24 weeks.
- Fasiglifam 50 mg: Fasiglifam 50 mg, tablets, orally, once daily, for up to 24 weeks.
Period: Overall Study
Arm/Group | Placebo | Fasiglifam 25 mg | Fasiglifam 50 mg
Started | 131 | 131 | 131
Completed | 55 | 58 | 59
Not Completed | 76 | 73 | 72
Not completed — Major Protocol Deviation | 1 | 0 | 0
Not completed — Adverse Event | 4 | 5 | 4
Not completed — Lost to Follow-up | 0 | 2 | 2
Not completed — Withdrawal by Subject | 6 | 4 | 0
Not completed — Study Termination | 64 | 61 | 65
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The randomized set included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Fasiglifam 25 mg | Fasiglifam 50 mg | Total
Number analyzed (Participants) | 131 | 131 | 131 | 393
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (12.41) | 55.1 (11.89) | 53.1 (10.96) | 53.6 (11.78)
Age, Customized [Number; unit: Participants]
  Less than (<) 65 years | 107 | 102 | 111 | 320
  Greater than or equal to (>=) 65 years | 24 | 29 | 20 | 73
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 61 | 44 | 169
  Male | 67 | 70 | 87 | 224
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 128 | 126 | 127 | 381
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 0 | 3
  White | 2 | 3 | 4 | 9
Body Mass Index [Mean (Standard Deviation); unit: Kilogram per square meter (kg/m^2)] | 26.00 (4.348) | 25.97 (3.989) | 26.12 (3.516) | 26.03 (3.956)
Smoking Classification [Number; unit: Participants]
  Never smoked | 89 | 90 | 71 | 250
  Current smoker | 31 | 16 | 33 | 80
  Ex-smoker | 11 | 25 | 27 | 63
Glycosylated Hemoglobin (HbA1c) Category [Number; unit: Participants]
  < 8.5 percent (%) | 98 | 99 | 107 | 304
  >= 8.5% | 33 | 32 | 24 | 89
Enrollment by Region [Number; unit: Participants]
  Australia | 6 | 5 | 6 | 17
  China | 70 | 70 | 70 | 210
  Korea, Republic of | 26 | 29 | 28 | 83
  New Zealand | 1 | 2 | 1 | 4
  Taiwan, Province of China | 28 | 25 | 26 | 79
Duration of Diabetes [Mean (Standard Deviation); unit: Years] — For this measure, number of participants evaluable were 125, 122, 124 for each arm respectively.
  Years | 2.293 (3.063) | 3.499 (3.64) | 2.182 (2.782) | 2.652 (3.227)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at Week 24
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Week 24 relative to baseline.
Time Frame: Baseline and Week 24
Population: Full Analysis Set (FAS) included of all randomized participants who received at least 1 dose of double blind study medication. Only participants with a baseline and at least 1 post-baseline value were included.
Measure: Least Squares Mean (Standard Error); unit: Percentage of Glycosylated Hemoglobin
Arm/Group | Placebo | Fasiglifam 25 mg | Fasiglifam 50 mg
Number analyzed (Participants) | 120 | 124 | 131
Percentage of Glycosylated Hemoglobin
  Baseline (n= 120, 124, 131) | 7.99 (0.104) | 7.94 (0.101) | 7.91 (0.102)
  Change at Week 24 (n= 52, 61, 59) | 0.15 (0.101) | -0.67 (0.097) | -0.87 (0.097)
Statistical Analysis 1: Comparison: Placebo vs Fasiglifam 50 mg; Assuming a standard deviation of 0.9% in change from baseline in HbA1c to Week 24 and a dropout rate of 15%, 210 participants per group provided at least 95% power to detect a treatment difference of 0.5% between treatment arms at a 2-sided significance level of 0.05; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures — Stepwise Comparison: 1) TAK-875 50 mg versus (vs.) placebo, 2) TAK-875 25 mg vs. placebo. Step 2 was performed only if p-value at step 1 was <=0.050; Treatment, country, visit, and visit-by-treatment interaction as fixed factors, baseline value as covariate; Least squares mean difference = -1.03, 95% CI 2-sided [-1.27 to -0.78], Standard Error of Mean 0.126
Statistical Analysis 2: Comparison: Placebo vs Fasiglifam 25 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Treatment, country, visit, and visit-by-treatment interaction as fixed factors, baseline value as covariate; Least squares mean difference = -0.82, 95% CI 2-sided [-1.07 to -0.57], Standard Error of Mean 0.126

2. Secondary Outcome: Percentage of Participants With HbA1c <7% at Week 24
Time Frame: Week 24
Population: FAS included of all randomized participants who received at least 1 dose of double blind study medication. Only Participants with a baseline and at least 1 post baseline value were included.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Fasiglifam 25 mg | Fasiglifam 50 mg
Number analyzed (Participants) | 120 | 124 | 131
Percentage of participants | 20.0 | 42.7 | 52.7
Statistical Analysis 1: Comparison: Placebo vs Fasiglifam 50 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic — No multiplicity adjustment; Treatment and baseline HbA1c as explanatory variables; Odds Ratio (OR) = 5.66, 95% CI 2-sided [2.99 to 10.72]
Statistical Analysis 2: Comparison: Placebo vs Fasiglifam 25 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic — No multiplicity adjustment; Treatment and baseline HbA1c as explanatory variables; Odds Ratio (OR) = 3.42, 95% CI 2-sided [1.81 to 6.49]

3. Secondary Outcome: Change in Fasting Plasma Glucose From Baseline to Week 24
Description: The change between the fasting plasma glucose value collected at Week 24 relative to baseline.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Milligram per deciliter (mg/dL)
Arm/Group | Placebo | Fasiglifam 25 mg | Fasiglifam 50 mg
Number analyzed (Participants) | 129 | 127 | 129
Milligram per deciliter (mg/dL)
  Baseline (n =129, 127, 129) | 152.4 (4.74) | 152.4 (4.67) | 149.7 (4.74)
  Change at Week 24 (n = 51, 58, 57) | 15.1 (3.59) | -20.6 (3.42) | -20.4 (3.45)
Statistical Analysis 1: Comparison: Placebo vs Fasiglifam 50 mg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures — No multiplicity adjustment; Treatment, country, visit, and visit-by-treatment interaction as fixed factors, baseline value covariate; Least squares mean difference = -35.6, 95% CI 2-sided [-44.2 to -26.9], Standard Error of Mean 4.36
Statistical Analysis 2: Comparison: Placebo vs Fasiglifam 25 mg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures — No multiplicity adjustment; Treatment, country, visit, and visit-by-treatment interaction as fixed factors, baseline value as covariate; Least Squares mean Difference = -35.7, 95% CI 2-sided [-44.3 to -27.1], Standard Error of Mean 4.36

4. Secondary Outcome: Change From Baseline in 2-hour Postprandial Glucose (PPG) Following Oral Glucose Tolerance Test (OGTT) at Week 24
Description: The change between the value of glucose after a meal, measured following OGTT collected at Week 24 relative to baseline. Oral glucose tolerance test measures glucose, insulin, and C-peptide through blood samples drawn at 0, 30, 60, 90, and 120 minutes following consumption of a 75 gram (g) glucose beverage.
Time Frame: Baseline and Week 24
Population: FAS included of all randomized participants who received at least 1 dose of double blind study medication. Only participants with a baseline and at least 1 post-baseline value were included.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Fasiglifam 25 mg | Fasiglifam 50 mg
Number analyzed (Participants) | 8 | 6 | 7
mg/dL
  Baseline | 150.3 (21.69) | 121.2 (22.76) | 129.0 (18.72)
  Change at Week 24 | 3.7 (24.58) | -21.2 (25.98) | 9.6 (21.15)
Statistical Analysis 1: Comparison: Placebo vs Fasiglifam 50 mg; Test type: Superiority or Other; p = 0.846, ANCOVA — No multiplicity adjustments; Treatment and country as fixed factors and baseline value as covariate; Least Squares Mean Difference = 5.9, 95% CI 2-sided [-57.9 to 69.6], Standard Error of Mean 29.72
Statistical Analysis 2: Comparison: Placebo vs Fasiglifam 25 mg; Test type: Superiority or Other; p = 0.427, ANCOVA — No multiplicity adjustments; Treatment and country as fixed factors and baseline value as covariate; Least Squares Mean Difference = -24.9, 95% CI 2-sided [-90.1 to 40.3], Standard Error of Mean 30.40

ADVERSE EVENTS:
Time Frame: Treatment -emergent adverse events are adverse events that started after the first dose of double- blind study drug and no more than 30 days after the last dose of double blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Fasiglifam 25 mg | Fasiglifam 50 mg
Serious Adverse Events (participants affected / at risk) | 5/131 | 5/131 | 8/131
Other Adverse Events (participants affected / at risk) | 39/131 | 51/131 | 50/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=131) | Fasiglifam 25 mg (N=131) | Fasiglifam 50 mg (N=131)
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Epiglottitis (Infections and infestations) | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=131) | Fasiglifam 25 mg (N=131) | Fasiglifam 50 mg (N=131)
Upper respiratory tract infection (Infections and infestations) | 8 | 6 | 8
Nasopharyngitis (Infections and infestations) | 5 | 10 | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 2 | 12
Dizziness (Nervous system disorders) | 5 | 7 | 2
Proteinuria (Renal and urinary disorders) | 3 | 5 | 5
Dyslipidaemia (Metabolism and nutrition disorders) | 3 | 4 | 5
Hyperlipidaemia (Metabolism and nutrition disorders) | 4 | 6 | 2
Blood creatine phosphokinase increased (Investigations) | 3 | 5 | 3
Headache (Nervous system disorders) | 2 | 4 | 3
Hypertension (Vascular disorders) | 1 | 4 | 3
Urinary tract infection (Infections and infestations) | 1 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 3 | 2
Insulin resistance (Metabolism and nutrition disorders) | 3 | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 3
Palpitations (Cardiac disorders) | 3 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 3
Chest pain (General disorders) | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.